CLINICAL TRIAL: NCT05944536
Title: The Effects of Single and Dual Task Balance Exercises in Substance Use Disorders: A Randomized Controlled Study
Brief Title: Single and Dual Task Balance Exercises in Substance Use Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara Yildirim Beyazıt University (Other)
Collaborators: Ankara Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022
Record Dates: First submitted 2023-07-06; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Substance Use Disorders
Keywords: Substance Abuse; Balance Exercise; Dual Task
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Patients who the inclusion criteria and agreed to participate were randomly allocates to Group 1 [Balance Exercises(BE)] and Group 2 [BE+Dual Tasks(DT)]
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balance Exercise (BE) (Active Comparator): Balance exercises; static standing on flat ground for 30 seconds, standing in tandem position for 30 seconds, standing on one foot for 30 seconds, standing on tiptoe for 30 seconds, looking left and right with one foot in the air, backward rotation with one foot in the air, rotation, squatting slightly in knee flexion with one foot in the air, squatting slightly in knee extension with one foot in the air, going on tiptoe and turning with the heel, multi-directional stretches on the balance board Each exercise will be performed with 10 repetitions for both lower extremities.
  Interventions: Other: Balance Exercises (BE)
- BE+Dual Task (Experimental): Cognitive and motor secondary tasks were given along with balance exercises. Cognitive tasks: color discrimination, counting city names, counting fruit and vegetable names, saying 3 numbers between 50-100, talking on a mobile phone, subtracting 3 and 7 in series, saying male names, counting backwards out loud, asking for a series of addition and subtraction operations.
  Motor tasks: carrying a glass of water, carrying a glass on a tray, carrying an object, pressing a button, transferring money from hand to hand, rhythmic clapping
  Interventions: Other: BE + Dual Task

INTERVENTIONS:
Other: Balance Exercises (BE) — Each exercise was performed with 10 repetitions for both lower limbs.
  Arms: Balance Exercise (BE)
Other: BE + Dual Task — Cognitive and motor secondary tasks were given
  Arms: BE+Dual Task

SUMMARY:
Changes in the brain reward pathway and brain tissue in alcohol and substance addiction cause balance disorders, cognitive problems, depression, and substance cravings in individuals. The aim of this study is to examine the effects of balance exercises and dual task balance exercises in individuals with alcohol or substance addiction who are receiving treatment.

DETAILED DESCRIPTION:
This randomized controlled trial was conduces in Ankara Training and Research Hospital, Alcohol and Substance Addiction Treatment Center, Turkey. Individuals who used substances for more than 1 year, between the ages of 18-50 and with a Mini-Mental State Examination score of 24 and above were included in the study. Individuals with orthopedic, neurological or systemic disease, problem with vision and hearing, a neurodevelopmental or neurocognitive disorder and active infection were excluded from the study. In addition, individuals under the effect of substances that negatively affect their cognitive functions were not included in the study. Before starting the study, the Mini-Mental State Examination was used to determine that the individuals were at a cognitive level to complete the tests to be applied. The demographic characteristics of the individuals were saved. The Stroop Test-Çapa Form was used to evaluate executive functions. Y Balance Test, Time Up Go Test and 10 meter walk test were used to evaluate balance. Patients were randomly divided into 2 groups. The first group received only balance exercise and the second group received balance exercise with motor and cognitive dual tasks.

ELIGIBILITY:
Inclusion Criteria:

* Being literate,
* Having a diagnosis of alcohol and substance use disorder according to The Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5),
* More than 1 year of substance abuse,
* Receiving treatment within the scope of the fight against addiction,
* Not participating in a regular exercise program in the last six months.

Exclusion Criteria:

* Scoring 23 and below on the Mini Mental Test,
* Having a neurodevelopmental or neurocognitive disorder,
* Being under the influence of drugs or alcohol in a way that negatively affects the person's -cognitive functions,
* Having a psychiatric disorder that requires treatment other than opiate and tobacco use disorder according to DSM-5 diagnostic criteria,
* Cognitive impairment due to mental retardation, drug/substance abuse or other medical condition that may cause difficulty in understanding the study instructions,
* Being diagnosed with any orthopedic, neurological and systemic disease,
* Having an active infection,
* Having problems with vision and hearing.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2023-07-15 (Estimated); Study Completion 2023-07-15 (Estimated)

PRIMARY OUTCOMES:
Dual Task Timing | 8 weeks
  the effect of dual tasks given alongside balance exercises on balance

CONTACTS AND LOCATIONS:
Overall Officials: Ertuğrul Demirdel, PhD, Study Director — Ankara Yildirim Beyazıt University; Beyza Gül Aşkın, MsC, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Yildirim Beyazit University, Faculty of Health Sciences, Department of Physical Therapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weiss NH, Gratz KL, Lavender JM. Factor Structure and Initial Validation of a Multidimensional Measure of Difficulties in the Regulation of Positive Emotions: The DERS-Positive. Behav Modif. 2015 May;39(3):431-53. doi: 10.1177/0145445514566504. Epub 2015 Jan 9. PMID 25576185
- [Background] Robertson CL, Ishibashi K, Chudzynski J, Mooney LJ, Rawson RA, Dolezal BA, Cooper CB, Brown AK, Mandelkern MA, London ED. Effect of Exercise Training on Striatal Dopamine D2/D3 Receptors in Methamphetamine Users during Behavioral Treatment. Neuropsychopharmacology. 2016 May;41(6):1629-36. doi: 10.1038/npp.2015.331. Epub 2015 Oct 27. PMID 26503310
- [Background] Colledge F, Vogel M, Dursteler-Macfarland K, Strom J, Schoen S, Puhse U, Gerber M. A pilot randomized trial of exercise as adjunct therapy in a heroin-assisted treatment setting. J Subst Abuse Treat. 2017 May;76:49-57. doi: 10.1016/j.jsat.2017.01.012. Epub 2017 Jan 29. PMID 28143679
- [Background] Wang D, Zhu T, Chen J, Lu Y, Zhou C, Chang YK. Acute Aerobic Exercise Ameliorates Cravings and Inhibitory Control in Heroin Addicts: Evidence From Event-Related Potentials and Frequency Bands. Front Psychol. 2020 Sep 29;11:561590. doi: 10.3389/fpsyg.2020.561590. eCollection 2020. PMID 33101132
- [Background] Gligoroska JP, Manchevska S. The effect of physical activity on cognition - physiological mechanisms. Mater Sociomed. 2012;24(3):198-202. doi: 10.5455/msm.2012.24.198-202. PMID 23678325
- [Background] Prasertsakul T, Kaimuk P, Chinjenpradit W, Limroongreungrat W, Charoensuk W. The effect of virtual reality-based balance training on motor learning and postural control in healthy adults: a randomized preliminary study. Biomed Eng Online. 2018 Sep 18;17(1):124. doi: 10.1186/s12938-018-0550-0. PMID 30227884
- [Background] Walaszek R, Chwala W, Walaszek K, Burdacki M, Blaszczuk J. Evaluation of the accuracy of the postural stability measurement with the Y-Balance Test based on the levels of the biomechanical parameters. Acta Bioeng Biomech. 2017;19(2):121-128. PMID 28869638
- [Background] Gungen C, Ertan T, Eker E, Yasar R, Engin F. [Reliability and validity of the standardized Mini Mental State Examination in the diagnosis of mild dementia in Turkish population]. Turk Psikiyatri Derg. 2002 Winter;13(4):273-81. Turkish. PMID 12794644
- [Background] Filipa A, Byrnes R, Paterno MV, Myer GD, Hewett TE. Neuromuscular training improves performance on the star excursion balance test in young female athletes. J Orthop Sports Phys Ther. 2010 Sep;40(9):551-8. doi: 10.2519/jospt.2010.3325. PMID 20710094
- [Background] MacLeod CM. Half a century of research on the Stroop effect: an integrative review. Psychol Bull. 1991 Mar;109(2):163-203. doi: 10.1037/0033-2909.109.2.163. No abstract available. PMID 2034749
- [Background] Sousa N, Sampaio J. Effects of progressive strength training on the performance of the Functional Reach Test and the Timed Get-Up-and-Go Test in an elderly population from the rural north of Portugal. Am J Hum Biol. 2005 Nov-Dec;17(6):746-51. doi: 10.1002/ajhb.20446. PMID 16254902
- [Background] Gribble PA, Hertel J, Plisky P. Using the Star Excursion Balance Test to assess dynamic postural-control deficits and outcomes in lower extremity injury: a literature and systematic review. J Athl Train. 2012 May-Jun;47(3):339-57. doi: 10.4085/1062-6050-47.3.08. PMID 22892416
- [Background] Sinaei, E., Kamali, F., Nematollahi, A., Etminan, Z. Comparing the effects of balance training with and without cognitive tasks on the quality of life and balance performance in community-dwelling older adults: a single-blind randomized clinical trial. Journal of Rehabilitation Sciences & Research, 2016; 3(4): 91-96. doi: 10.30476/jrsr.2016.41106
- See also: Clinical Assessment of Gait — https://doi.org/10.1016/B978-0-323-60913-5.00005-2